CLINICAL TRIAL: NCT07057765
Title: Predictive Value of CRP, Albumin, CAR, and mGPS in DLBCL: A Prospective Cohort Study on Treatment Outcomes and Toxicity
Brief Title: Predictive Value of CRP, Albumin, CAR, and mGPS in Treatment Outcomes of DLBCL
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD104/2025
Record Dates: First submitted 2025-06-02; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-05

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma; Markers of Inflammation
Keywords: DLBCL; CRP To Albumin Ratio; CAR; modified Glassgow Prognostic Score; mGPS
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with DLBCL Treated with R-CHOP (Observational Group): Patients diagnosed with diffuse large B-cell lymphoma (DLBCL) who are receiving R-CHOP chemotherapy as part of standard clinical care. This observational study aims to evaluate the predictive value of baseline inflammatory markers (CRP, albumin, CAR, and mGPS) on treatment response and toxicity. No study-specific interventions are administered.
  Interventions: Drug: Observational Assessment of Standard R-CHOP Treatment

INTERVENTIONS:
Drug: Observational Assessment of Standard R-CHOP Treatment — Patients will receive R-CHOP chemotherapy (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) as part of routine clinical care. The study does not assign or modify treatment. Data will be collected to assess the association between inflammatory markers and clinical outcomes.

SUMMARY:
This observational study evaluates the predictive value of systemic inflammatory markers-CRP, albumin, CRP-to-albumin ratio (CAR), and modified Glasgow Prognostic Score (mGPS)-in patients with diffuse large B-cell lymphoma (DLBCL) receiving R-CHOP chemotherapy. The study examines associations with treatment response, toxicity, and clinical characteristics.

DETAILED DESCRIPTION:
This prospective cohort study investigates the predictive significance of systemic inflammatory markers-CRP, serum albumin, CRP-to-albumin ratio (CAR), and modified Glasgow Prognostic Score (mGPS)-in patients with diffuse large B-cell lymphoma (DLBCL) treated with R-CHOP chemotherapy. The study aims to assess correlations between these markers and treatment outcomes, including objective response rate (ORR) and treatment-related toxicity. Inflammatory markers will be measured at baseline and after three chemotherapy cycles. Treatment response will be evaluated using Lugano classification criteria, and toxicity will be assessed per CTCAE version 5.0. The study also explores associations with clinical characteristics such as disease stage and performance status, aiming to enhance prognostic modeling and support personalized treatment strategies in DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 65 years
* Pathologically confirmed, treatment-naïve diffuse large B-cell lymphoma (DLBCL)
* Any stage of disease (nodal or extra-nodal), with or without B symptoms
* Scheduled to receive standard systemic treatment (R-CHOP)
* ECOG performance status 0-2
* Baseline normal:
* Complete blood count (CBC)
* Hepatitis viral markers
* Liver and renal function tests
* Urine analysis
* Echocardiogram
* Additional investigations to exclude current infection if clinically indicated

Exclusion Criteria:

* History of other concurrent or previous malignancies
* Relapsed or refractory DLBCL
* Uncontrolled comorbid conditions that may interfere with study participation, including:
* Diabetes mellitus
* Autoimmune diseases
* Active infections
* Chronic inflammatory diseases
* Cardiac dysfunction
* Liver cell failure
* Pregnant females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naïve, pathologically confirmed DLBCL patients who will attend the Clinical Oncology and Nuclear Medicine Department until the target sample size is reached. All participants will receive standard treatment protocol (R-CHOP) after providing informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Following 3 Cycles of R-CHOP Based on Baseline Inflammatory Markers | Baseline (Day 1 of Cycle 1) and Day 63 (End of Cycle 3; each cycle is 21 days)
  Proportion ( %) of patients achieving an objective response (complete or partial) according to the Lugano classification after three cycles of R-CHOP chemotherapy. Patients will be stratified by baseline inflammatory markers:
  * C-reactive protein (CRP, mg/L, measured by immunoturbidimetric assay)
  * Serum albumin (g/dL, measured by colorimetric assay)
  * CRP/Albumin ratio (CAR, calculated as CRP divided by albumin)
  * Modified Glasgow Prognostic Score (mGPS, range 0-2) Response will be assessed using PET/CT imaging.
Incidence of Treatment-Related Toxicity During Initial Treatment According to Baseline Inflammatory Markers | Day 1 of Cycle 1 through Day 63 (End of Cycle 3; each cycle is 21 days)
  Incidence (%) of patients experiencing any-grade treatment-related adverse events during the first three cycles of R-CHOP, stratified by baseline CRP, albumin, CAR, and mGPS. Toxicity will be graded according to CTCAE version 5.0.

SECONDARY OUTCOMES:
Proportion of Patients in Each IPI Risk Category by Baseline Inflammatory Marker Levels | Day 1 of Cycle 1 (each cycle is 21 days)
  Proportion (%) of patients in each International Prognostic Index (IPI) risk category (low, intermediate, high), stratified by baseline inflammatory markers:
  * CRP (mg/L, measured by immunoturbidimetric assay)
  * Albumin (g/dL, measured by colorimetric assay)
  * CRP/Albumin ratio (CAR, calculated as CRP divided by albumin)
  * Modified Glasgow Prognostic Score (mGPS, range 0-2) IPI will be calculated based on age, LDH level, Ann Arbor stage, ECOG performance status, and extranodal involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Ellithy, MD, Principal Investigator — Faculty of Medicine, Ain Shams University; Shaimaa A Pessar, MD, Study Director — Faculty of Medicine, Ain Shams University; Reham M Faheim, MD, Study Director — Faculty of Medicine, Ain Shams University; Doaa A Mohamed, MD, Study Director — Faculty of Medicine, Ain Shams University
Locations (1):
- Clinical Oncology and Nuclear Medicine Department, Faculty of Medicine, Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Because the study is conducted within an academic setting and involves patient data that cannot be shared publicly due to confidentiality and ethical considerations."